CLINICAL TRIAL: NCT04835519
Title: Open-Label, Nonramdominzed, Single-Arm Phase I/II Study to Evaluate the Safety and Tolerability of Functionally Enhanced CD33 CAR T Cells in Subjects With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Phase I/II Study of Enhanced CD33 CAR T Cells in Subjects With Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing Boren Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRYY-IIT-LCYJ-2021-003
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2023-02

CONDITIONS: Acute Myeloid Leukemia; Relapse Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chimeric antigen receptor T cell treatment (Experimental)
  Interventions: Biological: chimeric antigen receptor T cell

INTERVENTIONS:
Biological: chimeric antigen receptor T cell — Subjects will be pretreated with chemotherapy prior to infusion of CAR T cells: about 5 days before cells transfusion, the patients who planned to reinfuse CAR T cells were treated with fluorodarabine 30 mg/m^2( body surface area) and cyclophosphamide 250 mg/m^2( body surface area) for 3 days. Then this study will be using the Bayesian optimal interval phase I/II (Boin12) trial design. The protocol preset 2 dose levels: Dose 1 (DL-1) was 5×10^5 (±20%) CAR T cells/kg, and dose 2 (DL-2) was 1×10^6 (±20%) CAR T cells/kg. If the above dose cannot be met, subjects can still enter the study upon investigator consideration but require documentation of dosing. The lowest dose is 1×10^5 CAR T cells/kg (±20%), and the highest dose is 1×10^6 CAR T cells/kg (±20%). If the dose is out of the range mentioned above, entry into the trial will not be considered.

SUMMARY:
This is a open-label, nonramdominzed, single-arm, Phase I/II Study to evaluate safety and tolerability of functionally enhanced CD33 CAR-T cells in subjects with relapsed or refractory acute myeloid leukemia. 25 subjects will be enrolled. Subjects will be pretreated with chemotherapy prior to infusion of CAR T cells: about 5 days before cells transfusion, the patients who planned to reinfuse CAR T cells were treated with fluorodarabine 30 mg/m^2( body surface area) and cyclophosphamide 250 mg/m^2( body surface area) for 3 days. Then the Bayesian optimal interval phase I/II (Boin12) trial design will be used in this study: The protocol preset 2 dose levels: Dose 1 (DL-1) was 5×10^5 (±20%) CAR T cells/kg, and dose 2 (DL-2) was 1×10^6 (±20%) CAR T cells/kg. Phase I was the dose exploration phase. After determining the optimal biological dose (OBD), phase II will be expanded at the OBD dose by 10 cases, enrollment will reach 25 cases, and the trial will be discontinued. Moreover, the first 3 enrolled subjects per dose group will be on one by one dosing regimen.

The expected initial dose of 5×10^5 (±20%) CAR T cells/kg could not be achieved due to preparation problems and should be placed in the reduced dose group. The number of cells will be collected by the above regimen as far as possible. If this is not possible, subjects can still enter the study upon investigator consideration but require documentation of dosing. The lowest dose is 1×10^5 CAR T cells/kg (±20%), and the highest dose is 1×10^6 CAR T cells/kg (±20%). If the dose is out of the range mentioned above, entry into the trial will not be considered.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Candidates with relapse or refractory CD33+ acute myeloid leukemia, who have progressed on after treatment with all standard therapies or intolerant of standard care, have limited prognosis with currently available therapies and had no available curative treatment options (such as HSCT or chemotherapy)
2. Male or female, aged 1-70 years
3. No serious allergic constitution
4. Eastern Cooperative Oncology Group (ECOG) performance status (Oken et al.,1982) score 0 to 2
5. Have life expectancy of at least 60 days based on investigator's judgement
6. CD33 positive in bone marrow or cerebrospinal fluid (CSF) by flow cytometry, or CD33 positive in tumor tissues by immunohistochemistry; (CD33 positive criteria: Flow cytometry: Positive: > 80% of tumor cells expressed CD33 and the MFI of CD33 is the same as that in normal myeloid cells; Dim: > 80% of tumor cells expressed CD33, but the MFI of CD33 is lower than that in normal myeloid cells as least as 1log; Partial positive: 20-80% of tumor cells expressed CD33 and the MFI of CD33 is the same as that in normal myeloid cells. Tumor tissue immunohistochemistry: Positive > 30% tumor cells expressed CD33);
7. Provide a signed informed consent before any screening procedure; subjects who voluntarily participate in the study should have the ability to understand and sign the informed consent form and be willing to follow the study visit schedule and relevant study procedure, as specified in the protocol. Candidates aged 19-70 years need to be sufficiently conscious and able to sign the treatment consent form and voluntary consent form. Pediatric patients aged 1-7 years could be recruited after signing an informed consent form by a legal surrogate (Guardian); pediatric patients aged 8-18 years need to be sufficiently conscious and voluntarily signed an informed consent form, and their legal surrogates (guardians) were also required to sign a written informed consent form.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Intracranial hypertension or disorder of consciousness
2. Symptomatic heart failure or severe arrhythmia
3. Symptoms of severe respiratory failure
4. Complicated with other types of malignant tumors
5. Diffuse intravascular coagulation
6. Serum creatinine and / or blood urea nitrogen ≥ 1.5 times of the normal value
7. Suffering from septicemia or other uncontrollable infections
8. Patients with uncontrollable diabetes
9. Severe mental disorders
10. Obvious and active intracranial lesions were detected by cranial magnetic resonance imaging (MRI)
11. Have received organ transplantation (excluding hematopoietic stem cell transplantation);
12. Reproductive-aged female patients with positive blood HCG test
13. Screened to be positive of infection of hepatitis (including hepatitis B and C), AIDS or syphilis
14. Patients with tumor burden higher than 30% requiring reinfusion of autologous CAR-T cells.

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-05-19 (Actual)

PRIMARY OUTCOMES:
Incidence and type of dose-limiting toxicity (DLT) | day 21 post intravenous CAR T cell infusion
Incidence and severity of adverse events (AE) | day 28 post intravenous CAR T cell infusion

SECONDARY OUTCOMES:
CR (complete remission) rate and CRi (complete remission with incomplete blood count recovery) rate to the CAR-T treatment | day 15 post intravenous CAR T cell infusion
CR rate and CRi rate to the CAR-T treatment | day 28 post intravenous CAR T cell infusion

CONTACTS AND LOCATIONS:
Overall Officials: Jing Pan, MD/PhD, Principal Investigator — Beijing Boren Hospital
Locations (1):
- Beijing Boren Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No